CLINICAL TRIAL: NCT06789705
Title: Plasma Oxytocin Changes in Response to Low-dose MDMA vs. Placebo in Patients With Arginine Vasopressin Deficiency (Central Diabetes Insipidus) and Healthy Controls - the OxyMAX Study
Brief Title: Plasma Oxytocin Changes in Response to Low-dose MDMA vs. Placebo in Patients With Arginine Vasopressin Deficiency and Healthy Controls
Acronym: OxyMAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-01105; kt24ChristCrain3
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Central Diabetes Insipidus
Keywords: MDMA; oxytocin; arginin vasopressin
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Case-control study with a randomized, double-blind, controlled, cross-over design
Who Masked: Participant, Investigator
Masking Description: The order of the two MDMA doses is predefined in a randomization list. The randomization list is not known to the participants, the investigators and the study nurses involved in the trial. Participants and study personnel involved in supervising the session will be blinded to treatment order. The order is balanced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3,4-methylenedioxymethamphetamine (MDMA) and Placebo (Experimental): In this arm, first MDMA is given and after a wash-out phase of at least 10 days, Placebo will be administered.
  Interventions: Drug: MDMA; Other: Placebo
- Placebo and 3,4-methylenedioxymethamphetamine (MDMA) (Experimental): In this arm, first Placebo is given and after a wash-out phase of at least 10 days, MDMA will be administered.
  Interventions: Drug: MDMA; Other: Placebo

INTERVENTIONS:
Drug: MDMA — MDMA will be administered in a single dose of 50 mg (2 capsules of 25 mg MDMA) or 25mg (1 capsule of 25 mg MDMA, 1 capsule containing only mannitol filler) and given at treatment visit.
Other: Placebo — Placebo will be prepared as identical gelatin capsules containing only mannitol filler and given at treatment visit.

SUMMARY:
The investigator hypothesize that low-dose MDMA (3,4-methylenedioxymethamphetamine) will produce a sufficiently strong oxytocin stimulation in healthy controls and no relevant increase in patients. This study will confirm previously published data and provide important safety data with low-dose MDMA stimulation testing.

ELIGIBILITY:
Inclusion criteria patients:

1. Adult patients with confirmed diagnosis of Arginine Vasopressin deficiency (central diabetes insipidus)2 or with only anterior pituitary deficiency

Inclusion criteria healthy controls:

1. Adult healthy controls
2. Matched for age, sex, Body mass index, and oestrogen replacement/menopause/hormonal contraceptives to patients
3. No medication, except hormonal contraception

Exclusion Criteria:

1. Participation in a trial with investigational drugs within 30 days
2. Illicit substance use (except for cannabis) more than 10 times in lifetime or any time within the previous two months
3. Consumption of alcoholic beverages >15 drinks/week
4. Tobacco smoking >10 cigarettes/day
5. Cardiovascular disease (coronary artery disease, heart failure Left ventricular ejection fraction <40%, stroke in the last 3 months, atrial fibrillation/flatter, Wolff-Parkinson-White-Syndrome)
6. Uncontrolled arterial hypertension (>140/90 mmHg) or hypotension (<85mmHg)
7. Current or previous major psychiatric disorder (e.g., major depression, schizophrenia spectrum disorder)
8. Psychotic disorder in first-degree relatives
9. Regular intake of selective serotonin reuptake inhibitors or Monoamine oxidase inhibitors
10. Pregnancy and breastfeeding
11. Diagnosed Chronic Kidney Disease > grade III (glomerular filtration rate < 30ml/min)
12. Diagnosed liver cirrhosis or alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) levels 2.5 times above the normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve in plasma oxytocin level | up to 6 weeks
  Area under the concentration-time curve in plasma oxytocin level from baseline oxytocin measurement (before MDMA intake) to 5 hours after a single administration of 25 mg or 50 mg MDMA in patients with Arginine Vasopressin deficiency as compared to healthy controls.

SECONDARY OUTCOMES:
Peak change in oxytocin plasma level | up to 6 weeks
  Peak change in oxytocin plasma level assessed for MDMA and placebo between patients and healthy controls
Time course of plasma oxytocin levels | up to 6 weeks
  The outcome will be descriptive. The p-value for the treatment effect will be adjusted for multiple testing using the Bonferroni-Holm procedure.
  The time course of plasma and urine measures after intake of MDMA or placebo will be visualized by means of line plots and box-plots for patients and healthy controls.
Time course of plasma MDMA concentration | up to 6 weeks
  The outcome will be descriptive. The p-value for the treatment effect will be adjusted for multiple testing using the Bonferroni-Holm procedure.
  The time course of plasma and urine measures after intake of MDMA or placebo will be visualized by means of line plots and box-plots for patients and healthy controls.
Subjective/emotional effects assessed on numeric analogue scales (NASs) | up to 6 weeks
  NAS (e.g.,any drug effect, good drug effect, bad drug effect, trust, etc., 0-10) will be repeatedly used to assess subjective alterations in consciousness over time. NAS will be presented as a range from 0 to 10 marked with "not at all" on the left and "extremely" on the right. The following NAS will be used: "any effect", "good effect", "bad effect", "liking", "high", "happy", "fear", "stimulated", "feeling close to others", "concentration", "thinking", "open", "trust", "want to be with other people", "loss of sense of time", and "the boundaries between myself and my surroundings seemed to blur". Scales will be administered before and repeatedly after substance administration and will take 2 minutes to answer.
Recognition of emotions and body expressions in the Emotion from Body expression and Emotion from Face (EmBody/EmFace) task | up to 6 weeks
  The EmBody and EmFace subtasks comprise each of 42 stimuli showing body or facial expressions of angry, happy, or neutral affect. Stimuli last 1.5 seconds at 24 frames per second and are geometrically and optically standardized to prevent biases induced by ethnic cues (e.g., hair or skin tone) or clothing. The test is performed once during each treatment visit and 2-2.5 h after MDMA administration.
Recognition of emotions and body expressions in the face emotion recognition task (FERT) | up to 6 weeks
  At timepoint 150 min during the expected peak concentration of MDMA participants will perform FERT. The FERT is used to assess recognition of basic emotions. The task includes 10 neutral faces and 160 faces that express one of four basic emotions (i.e., happiness, sadness, anger, and fear), with pictures morphed between 0% (neutral) and 100% in 10% steps. Two female and two male pictures are used for each of the four emotions.
Anxiety level with the State-Trait Anxiety Inventory (STAI-S) | up to 6 weeks
  Anxiety level assessed for MDMA and placebo between patients and healthy controls with STAI.
  The state score (STAI-S) evaluates the current state of anxiety, asking how respondents feel "right now," using items that measure subjective feelings of apprehension, tension, nervousness, worry, and activation/arousal of the autonomic nervous system.
  Based on responses to 20 items, with scores ranging from 1 ("almost never") to 4 ("almost always"), a total score is calculated. The total trait score (STAI-T) ranges from 20 to 80, with higher scores indicating more pronounced anxiety and scores. The state score (STAI-S) evaluates the current state of anxiety, asking how respondents feel "right now," using items that measure subjective feelings of apprehension, tension, nervousness, worry, and activation/arousal of the autonomic nervous system.
Anxiety level with the State-Trait Anxiety Inventory (STAI-T) | at baseline
  Anxiety level assessed for MDMA and placebo between patients and healthy controls with STAI.
  This is a questionnaire given to adults to determine the general anxiety levels. Based on responses to 20 items, with scores ranging from 1 ("almost never") to 4 ("almost always"), a total score is calculated. The total trait score (STAI-T) ranges from 20 to 80, with higher scores indicating more pronounced anxiety and scores.The STAI-T evaluates relatively stable aspects of "anxiety proneness," including general states of calmness, confidence, and security. A score above 45/80 indicating clinically significant anxiety symptoms.
Number of complaints | up to 6 weeks
  Documenting list of complaints (LC)
Number of adverse effects | up to 6 weeks
  Documenting all adverse effects
Time course of plasma copeptin | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Time course of plasma Adrenocorticotropic hormone (ACTH) | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Time course of plasma cortisol | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Time course of plasma prolactin | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Time course of plasma neurophysin I | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Alexithymia level using the Toronto-Alexithymia-Scale 20 (TAS-20) | up to 6 weeks
  Alexithymia is described as a trait to identify and describe emotions experienced by oneself or others. It is characterized by a marked difficulty in consciously experiencing, identifying, and describing emotions, as well as reduced introspection. The TAS 20 has a three-factor structure: Difficulty identifying feelings, difficulty describing feelings and externally oriented thinking. It includes 20 questions with scores ranging from 1 (strongly disagree) to 5 (strongly agree).
Depression level using the Beck-Depressions-Inventory II (BDI-II) | up to 6 weeks
  The BDI II is one of the most used self-reported scales for measuring depression. It uses 21 items ranked from 0 (symptom absent) to 3 (severe symptoms) to measure the severity of depression.
  The self-administered form takes about 5-10 minutes for the participant. The minimum score is 0 and maximum score is 63. In non-clinical populations, scores above 20 indicate depression. In those diagnosed with depression, scores of 0-13 indicate minimal depression, 14-19 (mild depression), 20-28 (moderate depression) and 29-63 (severe depression).
General physical & mental health using the posterior-pituitary quality of life questionnaire (PP-QoL) | up to 6 weeks
  PROMIS measures are relevant across all conditions to assess clinical symptoms, functioning, and quality of life. This questionnaire will consist of 29 items. In addition, cognitive functions consisting of 4 items and sociodemographic core data will be asked. PROMIS measures have been developed and validated with state-of-the-science methods to be psychometrically sound and to transform how life domains are measured. They have greater precision than most conventional measures. Greater precision (less error) enhances power in a less costly way than increasing sample size. PROMIS measures are relevant across all conditions to assess clinical symptoms, functioning, and quality of life.
General physical & mental health using the Patient-Reported Outcomes Measurement Information System (PROMIS) | up to 6 weeks
  The PROMIS is a set of person-centred measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS measures can be used with the general population and with individuals living with chronic conditions.PROMIS measures are relevant across all conditions to assess clinical symptoms, functioning, and quality of life. This questionnaire will consist of 29 items. In addition, cognitive functions consisting of 4 items and sociodemographic core data will be asked. PROMIS measures have been developed and validated with state-of-the-science methods to be psychometrically sound and to transform how life domains are measured. They have greater precision than most conventional measures. Greater precision (less error) enhances power in a less costly way than increasing sample size. PROMIS measures are relevant across all conditions to assess clinical symptoms, functioning, and quality of life.
Autistic traits level using the Autism-Spectrum Quotient Test (AQ) | up to 6 weeks
  This questionnaire is a diagnostic test designed to measure the expression of Autism Spectrum Disorder (ASD) traits in an individual by his or her subjective self-assessment. The AQ consists of 50 items, with four choices for each item from "definitely agree" to "definitely disagree" and a total score from 0 to 50. A score above the proposed cut-off of 29 highlights significant traits of autism.
Eating disturbances level using the Three-Factor Eating Questionnaire-Revised 18 Item (TFEQ-R18) | up to 6 weeks
  The TFEQ-R18 developed by Karlsson et al.118, assesses three dimensions of eating behavior: cognitive restraint, uncontrolled eating, and emotional eating. It consists of 18 items rated on a 4- point Likert scale and includes six items for cognitive restraint, nine for uncontrolled eating, and three for emotional eating. Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating. The reliability of each scale was computed using Cronbach's alphas. The overall reliability was acceptable (Cronbach's alpha = 0.82).
Resting energy expenditure (REE) in kcal per 24 hours, time course of plasma glucose, insulin and c-peptide, subjective saturation effects assessed on a 10-point NAS. | up to 6 weeks
  Indirect calorimetry for measurement of REE will be assessed after the expected plasma peak concentration of MDMA at 180min. Participant will be in an air-conditioned room with a room temperature between 22-24° C and wearing light clothing. To avoid activation of cold-induced thermogenesis and ensure a comfortably warm body surface temperature the patient will be covered by a blanket during the measurement of REE. Energy expenditure will then be measured with the ventilated hood technique using a Cosmed Quark Resting metabolic rate (RMR) for 30 minutes. Furthermore, participants will be asked to only perform a maximum of 30 minutes of medium exercise during the preceding 24 h.The unit of REE is kcal per 24 hours. It is assessed by volume of oxygen uptake (VO2) and expelled volume of carbon dioxide (VO2) in ml/min and calculated by the Weir Equation REE = [3.9 * (VO2) + 1.1 (VCO2)] * 1.44. The respiratory quotient (RQ) is calculated by dividing VCO2 by VO2.
Time course of plasma glucose | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Time course of plasma insulin | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Time course of plasma c-peptide | up to 6 weeks
  Samples will be taken for analysis and collected during the study days
Subjective saturation effects | up to 6 weeks
  Assessed on a 10-point Numeric Analog Scale (NAS). NAS will be presented as a range from 0 to 10 marked with "not at all" on the left and "extremely" on the right. The following NAS will be used: "any effect", "good effect", "bad effect", "liking", "high", "happy", "fear", "stimulated", "feeling close to others", "concentration", "thinking", "open", "trust", "want to be with other people", "loss of sense of time", and "the boundaries between myself and my surroundings seemed to blur".
Assessments of clinical variable blood pressure | up to 6 weeks
  Assessment of blood pressure
Assessments of clinical variable heart rate | up to 6 weeks
  Assessment of heart rate
Assessments of clinical variable body temperature | up to 6 weeks
  Assessment of body temperature
Assessments of laboratory variable plasma sodium | up to 6 weeks
  Assessment of plasma sodium
Assessments of laboratory variable potassium | up to 6 weeks
  Assessment of potassium

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland